CLINICAL TRIAL: NCT01243528
Title: Prospective, Non-interventional Observational Study at the Influence of Malnutrition on Nosocomial Infections in Patients During Early Neurological Rehabilitation
Brief Title: Observational Study at the Influence of Malnutrition on Infections
Acronym: Malnutrition
Status: Completed | Type: Observational
Sponsor: Marion Mertl-Roetzer (Other)
Responsible Party: Sponsor-Investigator, Marion Mertl-Roetzer, Head Physician, Schoen Clinic Bad Aibling
Organization: Schoen Clinic Bad Aibling (Other)
Other Study IDs: PINI01
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Malnutrition
Keywords: Malnutrition; Infection; Neurological
MeSH Terms: conditions — Malnutrition; Infections; Neurologic Manifestations | interventions — Laboratory Critical Values; Vitamin D; Creatinine; Blood Urea Nitrogen; Albumins; Prealbumin; Proteins; C-Reactive Protein; Triiodothyronine; Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in neurological rehabilitation: Patients suffering from a neurological disease
  Interventions: Other: Laboratory values

INTERVENTIONS:
Other: Laboratory values — Laboratory values which represent nutritional status
  Other Names: Vitamin D; Creatinine; Urea nitrogen; Albumin; Prealbumin; Total protein; C-reactive protein; Triiodothyronine; Thyroxin

SUMMARY:
The purpose of this trial is to determine whether nutritional status has an impact on nosocomial infections. Study population are patients undergoing early neurological rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in early neurological rehabilitation
* informed consent given

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in neurological rehabilitation facility
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 8 weeks
  Nutritional status is represented by Prognostic Inflammatory and Nutritional Index Score (PINI) and bioimpedanz-anlaysis-measurement (BIA)

SECONDARY OUTCOMES:
Nosocomial infections | 8 weeks
  Survey whether the patient has infections during the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Marion Mertl-Rötzer, Dr. med., Principal Investigator — Schoen Clinic Bad Aibling
Locations (1):
- Schoen Clinic Bad Aibling, Bad Aibling, Bavaria, Germany